CLINICAL TRIAL: NCT04013321
Title: Naturalistic Monitoring and Treatment of Chronic Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Devon Hansen, Assistant Professor, Washington State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 17379-002; KL2TR002317 (NIH)
Record Dates: First submitted 2019-06-17; First posted 2019-07-09 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Test intervention group (Experimental): Chronic insomniacs will track their sleep with the SleepScore Max device and will receive feedback and coaching from the Smartphone app associated with the device.
  Interventions: Device: SleepScore Max coaching feature
- Active control (Active Comparator): Chronic insomniacs in the active control group will be tracking their sleep with the device, without feedback or coaching. But they will also undergo online cognitive behavioral therapy for insomnia (CBTi).
  Interventions: Behavioral: Online CBTi
- Passive control (No Intervention): Chronic insomniacs in the passive control group will track their sleep using the SleepScore Max device, but without the feedback or coaching feature.
- Healthy control (No Intervention): Healthy sleepers will track their sleep using the SleepScore Max device, but without the feedback or coaching feature.

INTERVENTIONS:
Device: SleepScore Max coaching feature — The SleepScore max is a non-contact sleep tracking device. The app has an integrated feedback coaching feature to improve sleep.
  Arms: Test intervention group
Behavioral: Online CBTi — Online Cognitive Behavioral Therapy for insomnia is a user guided program to track sleep, receive sleep coaching, and initiate behavioral techniques such as tailored sleep scheduling and sleep hygiene to help improve sleep.
  Arms: Active control

SUMMARY:
90 individuals with chronic insomniacs and 30 healthy normal sleepers will have their sleep monitored by the SleepScore Max for 10 weeks. Individuals with chronic insomnia will be randomized into one of three groups (30 subjects in each): a test intervention group, a passive control group, and an active control group. The purpose of the study is to examine if the SleepScore max provides a accurate measurement of sleep relative to a validated, wrist-worn sleep monitor and if a integrated coaching feature within the SleepScore Max facilitates improvement in sleep relative to other gold standard treatment methods.

DETAILED DESCRIPTION:
90 chronic insomniacs, carefully screened using the criteria of Chronic Insomnia Disorder according to the International Classification of Sleep Disorders 3 (ICSD-3), will be studied. Additionally, 30 healthy normal sleepers will be included as controls. The duration of study participation will be 10 weeks. All subjects will wear an actigraph during week 1 to record baseline sleep patterns, followed by 8 weeks of recording with the SleepScore Max. During week 10, the subjects will wear the actigraph again to measure post intervention sleep. The healthy subjects will be used as a control to test if the SleepScore Max can track sleep well as compared to actigraphy. The subjects with chronic insomnia will be randomized into one of three groups (30 subjects in each). One of these groups is the test intervention group, in which subjects will track their sleep with the SleepScore Max device and will receive feedback and coaching from the Smartphone app associated with the device. The other two groups will serve as passive and active controls. The passive control group will track their sleep using the SleepScore Max device, but without any feedback or coaching. The active control group will also be tracking their sleep with the device, without feedback or coaching, but they will also undergo online CBTi which is a user guided program to track sleep, receive sleep coaching, and initiate behavioral techniques such as tailored sleep scheduling and sleep hygiene to help improve sleep.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Physically and psychologically healthy (except for chronic insomnia for the insomnia participants) as assessed by questionnaires and history
* No sleep disorders other than chronic insomnia (for insomnia participants only) as assessed by questionnaires and history
* Has daily access to an iPhone

Exclusion Criteria:

* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Sleep Duration | 10 weeks
  Quantify sleep duration using SleepScore Max in:
  * Passive control insomniacs vs healthy controls
  * Insomnia groups
Sleep Duration | 10 weeks
  Quantify sleep duration using Actigraphy in:
  * Passive control insomniacs vs healthy controls
  * Insomnia groups

SECONDARY OUTCOMES:
Sleep latency | 10 weeks
  Quantify sleep latency using SleepScore Max in:
  * Passive control insomniacs vs healthy controls
  * Insomnia groups
Sleep latency | 10 weeks
  Quantify sleep latency using actigraphy in:
  * Passive control insomniacs vs healthy controls
  * Insomnia groups
Intermittent wakefulness | 10 weeks
  Quantify intermittent wakefulness using SleepScore Max in:
  * Passive control insomniacs vs healthy controls
  * Insomnia groups
Intermittent wakefulness | 10 weeks
  Quantify intermittent wakefulness using actigraphy in:
  * Passive control insomniacs vs healthy controls
  * Insomnia groups

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep and Performance Research Center, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No
pending